CLINICAL TRIAL: NCT03261843
Title: The Effect of Using Autologous Platelet Rich Plasma on Posterior Lumbar Interbody Fusion : a Randomized Comparative Trial
Brief Title: The Effect of Using Autologous Platelet Rich Plasma on Posterior Lumbar Interbody Fusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelazim Abdelrahim Hassan, resident of orthopedics and trauma surgery, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: platelet rich plasma
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Autologous Platelet Rich Plasma Effect on Bone Healing
Keywords: platelet rich plasma , posterior lumbar interbody fusion

STUDY DESIGN:
Intervention Model Description: single center, prospective randomized comparative trial
Who Masked: Outcomes Assessor
Masking Description: the person performing the statistical analysis shall be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- posterior lumbar interbody fusion + platelet rich plasma (Active Comparator): the addition of autologous platelet rich plasma to the bone graft
  Interventions: Biological: autologous platelet rich plasma
- posterior lumbar interbody fusion (Active Comparator): bone graft alone
  Interventions: Procedure: posterior lumbar interbody fusion without autologous platelet rich plasma

INTERVENTIONS:
Biological: autologous platelet rich plasma — adding autologous platelet rich plasma to the bone graft harvested from the patient
  Arms: posterior lumbar interbody fusion + platelet rich plasma
Procedure: posterior lumbar interbody fusion without autologous platelet rich plasma — performing posterior lumbar interbody fusion without using platelet rich plasma
  Arms: posterior lumbar interbody fusion

SUMMARY:
the study aims to determine the effect of using Autologous platelet rich plasma on both the quality & rate of posterior lumbar interbody fusion & its outcome on the Patient regarding postoperative lumbar pain & functional outcome

DETAILED DESCRIPTION:
The study will be submitted for approval by the Ethics Committee of Faculty of Medicine, Assiut University, and written informed consent will be obtained from all patients prior to enrollment. The study population will be selected from patients attending the Department of Orthopedics and Trauma surgery, Assiut University hospitals.

Sixty patients will be selected for the study and will be randomized into two group one receiving posterior lumbar interbody fusion with Autologous platelet rich plasma and the other group will receive posterior lumbar interbody fusion without Autologous platelet rich plasma.

Methodology pre-operative preparation: Prior to the operation the selected patients will perform lumbar spine Computarised tomography and X ray films. Both the visual analogue scale of pain and the Oswestry disability index will be collected from the patients

Autologous platelet rich plasma preparation:

Autologous Platelet rich plasma is obtained using a two-stage centrifugation process.

Whole blood sample will be drawn from the participant and be collected in a sterile tube containing anticoagulant (sodium citrate 3.8% or Ethylenediaminetetraacetic acid ). The tube will be centrifuged at 160xg relative centrifugal force (about 1000 round per minute) for 10 min in a centrifugal apparatus. The first spin will separate platelet poor plasma at the top from red blood cells at the bottom and platelet rich plasma above (mixed with the white blood cells in the buffy coat). The Platelet poor plasma, Platelet rich plasma and a few red blood cells will be aspirated into a new tube, mixed and in the second spin, the tube will be centrifuged at 400xg relative centrifugal form (about 1500 round per minute) for another 10 minutes. The upper section will consist of Platelet poor plasma and the Platelet rich plasma will be collected at the bottom of the tube in the form of pellet. Then, Platelet poor plasma and Platelet rich plasma will be aspirated and mixed (discarding the upper portion). Prior to treatment calcium chloride 3% will be added to activate platelets immediately before its application to avoid coagulation of the specimen (for every 1.5 milliliter plasma, 1 milliliter calcium chloride 3% is added).

Surgery:

A posterior lumbar interbody fusion with posterior pedicle screw fixation will be performed through a midline posterior approach. Trans-pedicular screws will be placed under fluoroscopic guidance, followed by discectomy. The vertebral body endplates will be prepared by curetting until point bleeding was seen.

Autologous cancellous bone chips will be harvested unilaterally from the iliac wing, approached through the midline posterior incision. The bone chips will be steeped in the plasma solution until clotting occurred visually (approximately 10 minutes). In the control group, the bone chips will be filled with autologous bone in the same way and were implanted after approximately 10 minutes without incubation in a plasma solution.

ELIGIBILITY:
Inclusion Criteria:

* Spondylolisthesis.
* Degenerative disc disease requiring posterior lumbar interbody fusion not responding to medical treatment for 1 year.
* Age between 20 & 70 years.
* Single or multiple level fusions.

Exclusion Criteria:

* Previous lumbar spine surgery.
* Other lumbar spine pathology
* severe osteoporosis
* Chronic use of steroid or non-steroidal anti-inflammatory drugs (more than one year)
* Patients younger than 20 years old.
* Patients older than 70 years old.
* Immunocompromised patients (eg. Chronic renal failure)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
bridging trabecular bone scale | from 3 to 6 month post-operative
  the degree of bridging bone across the fused vertebral bodies

SECONDARY OUTCOMES:
visual analogue of pain | from 3 to 6 month post-operative
  the amount of pain sensed by the patient pre and post-operative
the Oswestry disability index | from 3 to 6 month post-operative
  the functional outcome on the patient

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Smith PA. Intra-articular Autologous Conditioned Plasma Injections Provide Safe and Efficacious Treatment for Knee Osteoarthritis: An FDA-Sanctioned, Randomized, Double-blind, Placebo-controlled Clinical Trial. Am J Sports Med. 2016 Apr;44(4):884-91. doi: 10.1177/0363546515624678. Epub 2016 Feb 1. PMID 26831629
- [Result] Sys J, Weyler J, Van Der Zijden T, Parizel P, Michielsen J. Platelet-rich plasma in mono-segmental posterior lumbar interbody fusion. Eur Spine J. 2011 Oct;20(10):1650-7. doi: 10.1007/s00586-011-1897-0. Epub 2011 Jul 10. PMID 21744284
- [Result] Weiner BK, Walker M. Efficacy of autologous growth factors in lumbar intertransverse fusions. Spine (Phila Pa 1976). 2003 Sep 1;28(17):1968-70; discussion 1971. doi: 10.1097/01.BRS.0000083141.02027.48. PMID 12973143
- [Result] Hee HT, Majd ME, Holt RT, Myers L. Do autologous growth factors enhance transforaminal lumbar interbody fusion? Eur Spine J. 2003 Aug;12(4):400-7. doi: 10.1007/s00586-003-0548-5. Epub 2003 May 22. PMID 12761669
- [Result] Kaux JF, Le Goff C, Seidel L, Peters P, Gothot A, Albert A, Crielaard JM. [Comparative study of five techniques of preparation of platelet-rich plasma]. Pathol Biol (Paris). 2011 Jun;59(3):157-60. doi: 10.1016/j.patbio.2009.04.007. Epub 2009 May 28. French. PMID 19481375
- [Result] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519
- [Result] Ferrari M, Zia S, Valbonesi M, Henriquet F, Venere G, Spagnolo S, Grasso MA, Panzani I. A new technique for hemodilution, preparation of autologous platelet-rich plasma and intraoperative blood salvage in cardiac surgery. Int J Artif Organs. 1987 Jan;10(1):47-50. PMID 3570542